CLINICAL TRIAL: NCT07027800
Title: Effects of High-intensity Resistance Training and Creatine Supplementation on Muscle Quality and Cognition in Perimenopausal Women: a Pilot Study
Brief Title: High Intensity Resistance Training + Creatine in Perimenopause
Acronym: PERIHIRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 24-3202
Record Dates: First submitted 2025-06-02; First posted 2025-06-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Perimenopause
Keywords: resistance training; muscle mass; hormone health; creatine monohydrate; exercise; nutrition; womens health
MeSH Terms: conditions — Motor Activity | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Creatine Monohydrate (Experimental): 20 g Creatine Monohydrate for 5 days followed by 5 grams creatine monohdyrate daily + 2 x weekly high intensity resistance training
  Interventions: Dietary Supplement: Creatine Monohydrate
- Placebo (Placebo Comparator): 20 g Non-Caloric Placebo followed by 5 grams daily placebo + 2 x weekly high intensity resistance training
  Interventions: Dietary Supplement: Placebo
- Control (No Intervention): No exercise or supplement provided

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — 20 gram loading of creatine monohdyrate for 5 days, followed by 5 grams per day for 6 weeks
  Arms: Creatine Monohydrate
Dietary Supplement: Placebo — 20 grams daily of non-caloric placebo + 5 grams daily non-caloric placebo for 6 weeks
  Arms: Placebo

SUMMARY:
Purpose: The aims of the study are to investigate the effects of high-intensity resistance training (HIRT) with or without creatine monohydrate (CM) supplementation on three key areas: muscle characteristics, brain health, and metabolism/protein dynamics.

Participants: 51 healthy, perimenopausal women between 38-60 years old. Procedures: In a randomized double-blind, placebo-controlled design, participants will either consume creatine (CM), a placebo (PL), or no supplement (CON). CM and PL groups will be assigned a HIRT protocol, and the CON will do no training.

DETAILED DESCRIPTION:
Over one million women in the U.S. transition through menopause each year, a phase marked by significant hormonal fluctuations (estrogen, progesterone, luteinizing hormone) and associated with increased cardiometabolic and cardiovascular risks. Research from our lab has identified key metabolic disruptions during the perimenopausal (PERI) period, including reduced protein balance, increased abdominal fat, decreased strength, and impaired metabolic flexibility. Additionally, women as early as age 35 may experience menopause-related symptoms such as cognitive decline, mood disturbances, and sleep disruptions.

Skeletal muscle health, critical for lifelong function, often begins to decline during PERI. While resistance training is known to improve muscle strength and body composition in older women, limited research has focused specifically on the PERI stage. High-intensity resistance training (HIRT) offers a time-efficient strategy to address these issues. Creatine monohydrate (CM) supplementation, traditionally used to enhance muscle performance, has shown potential benefits for cognitive function, mood, fatigue reduction, and overall metabolic health-effects particularly relevant to PERI women.

This pilot study aims to evaluate the preliminary effects of six weeks of HIRT, with or without CM supplementation, on muscle characteristics, brain health, and metabolism in women around PERI age. The study uses a randomized, double-blind, placebo-controlled design with broad inclusion criteria to enhance generalizability. Participants will undergo a 5-day supplementation phase followed by a 6-week training phase. Outcomes will include assessments of muscle quality and strength, cognitive function, brain oxygenation, metabolic rate, and protein turnover, while accounting for hormonal fluctuations.

This trial will provide foundational data to inform a larger, more comprehensive study and aims to identify effective, accessible interventions to support health and quality of life in women during the menopause transition.

ELIGIBILITY:
Inclusion Criteria:

* Women transitioning through perimenopause (defined by the North American Menopause Society Menopause Health Questionnaire), with or without hormone therapy or experiencing two or more perimenopause-related symptoms, as determined from the validated North American Menopause Society
* Women ≥38-60 yrs.
* Recreationally active [(≥30 minutes of moderate-intensity physical activity per week and <3 times per week of progressive resistance training, as defined by the International Physical Activity Questionnaire (IPAQ)]
* Body mass index of 18.5-34.9 kg/m^2
* Is at risk or has a current chronic disease that is not contraindicated by exercise, and could be improved by resistance exercise (i.e. type 2 diabetes, heart disease, hypertension, hypercholesterolemia, hyperthyroidism, depression, osteoporosis, etc.)

Exclusion Criteria:

* Experienced a musculoskeletal injury within the past three months that inhibits participation in the study.
* Has chronic kidney disease, liver disease, chronic obstructive pulmonary disease, or cancer
* Currently using medications that may directly impact the primary outcomes including: diuretics and corticosteroids).
* Currently using creatine monohydrate or other performance-enhancing supplements
* Has a self-identified or clinically diagnosed eating disorder
* Currently pregnant or planning to become pregnant (determined from urine pregnancy test)
* Currently nursing or have had a child within the previous 6 months
* Has participated in another clinical trial within four weeks prior to enrollment that in the opinion of the PI would influence the results.
* Has severely impaired hearing or speech or inability to speak English.
* Unwilling or unable to comply with the study protocol, including abstaining from caffeine, tobacco, alcohol, and physical activity before testing days.

Ages: 38 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 51 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Muscle quality | Baseline to after 6 weeks of resistance training and supplementation
  Muscle quality measured by echo intensity via ultrasound
Muscle Strength | Baseline to post 6 weeks of resistance training and supplementation
  Maximal strength from 1 repetition maximum for leg press

SECONDARY OUTCOMES:
Menopausal Symptoms | Baseline to post 6 weeks of resistance training + supplementation
  Greene climacteric Scale, 21 questions, scores ranging from 0-63, with higher number indicating greater symptom severity.
Resting metabolic rate | Baseline to post 6 weeks of resistance training + supplementation
  Resting metabolic rate determined from indirect calorimetry
Inventory of Depression and Anxiety | Baseline to post 6 weeks of resistance training + supplementation
  Inventory of Depression and Anxiety Symptoms (IDAS) questionnaire is based on a 5-point Likert scale, ranging from 'not at all' to 'extremely', scores ranging 0-63, with a higher score indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carollina at Chapel Hill
Locations (1):
- Applied Physiology Laboratory, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
This is pilot data and therefore may not be powered for secondary analyses